CLINICAL TRIAL: NCT04339777
Title: A Phase II Study of Allogeneic Hematopoietic Stem Cell Transplant for Patients With Inborn Errors of Immunity
Brief Title: Allogeneic Hematopoietic Stem Cell Transplant for Patients With Inborn Errors of Immunity
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200070; 20-C-0070
Record Dates: First submitted 2020-04-08; First posted 2020-04-09 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09-11

CONDITIONS: Lymphoproliferative Disorders; Autoimmune Lymphoproliferative; Immune System Diseases; Common Variable Immunodeficiency; Primary T-cell Immunodeficiency Disorders
Keywords: Autoimmunity; Haploidentical; Opportunistic Infection; Immune Dysregulation; Congenital
MeSH Terms: conditions — Lymphoproliferative Disorders; Immune System Diseases; Common Variable Immunodeficiency; T cell immunodeficiency primary; Autoimmune Diseases; Opportunistic Infections | interventions — fludarabine; Busulfan; Alemtuzumab; Whole-Body Irradiation; Tacrolimus; Mycophenolic Acid; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Low Intensity, Intermediate Intensity and High Intensity Conditioning with or without alemtuzumab
  Interventions: Drug: Busulfan test dose; Drug: Fludarabine; Drug: Busulfan; Drug: Alemtuzumab; Procedure: Allogeneic HSCT; Drug: Tacrolimus (Tacro); Drug: Mycophenolate mofetil (MMF); Drug: Cyclophosphamide (Cytoxan)
- Arm B (Active Comparator): Intermediate Intensity Conditioning with or without Alemtuzumab
  Interventions: Drug: Busulfan test dose; Drug: Fludarabine; Drug: Busulfan; Drug: Alemtuzumab; Radiation: Total body Irradiation; Procedure: Allogeneic HSCT; Drug: Tacrolimus (Tacro); Drug: Mycophenolate mofetil (MMF); Drug: Cyclophosphamide (Cytoxan)

INTERVENTIONS:
Drug: Busulfan test dose — 0.8 mg/kg IV infusion over 2 hours
Drug: Fludarabine — 40 mg/m2 IV infusion over 30 min once daily for 4 days
Drug: Busulfan — AUC Targeted Dose based on busulfan test dose PKs, IV infusion over 3 hours once daily (3.2 mg/kg IV per day will be the default dose) per the below time frame: For 10/10 Matched Related and Unrelated Donor Recipients For the High Intensity Arm, the busulfan dose will be given for 4 days (-6, -5, -4, and -3).
  For Intermediate Intensity Arm, the busulfan dose will be given for 3 days (-6,-5, and -4).
  For Low Intensity Arm, the busulfan dose will be given for 2 days on days (-6 and -5). 9/10 HLA Matched Related or Unrelated Donor Recipients For the High Intensity Arm, the busulfan dose will be given for 3 days (-6,
  -5, and -4). For the the Intermediate Intensity Arm, the busulfan dose will be given for 2 days (-6 and -5).
  For the Low Intensity Arm, the busulfan dose will be given for 1 day on day (-6).
Drug: Alemtuzumab — Alemtuzumab will be given if there is evidence of immune dysregulation 10 mg/m2 SC divided over three days (-14, -13, and -12)
Radiation: Total body Irradiation — 200 cGy Transplant Day -1 (Only for 9/10 HLA Matched Related or Unrelated Donor Recipients )
  Arms: Arm B
Procedure: Allogeneic HSCT — Stem cell transplant
Drug: Tacrolimus (Tacro) — Tacrolimus 0.02 mg/kg IV continuous infusion over 24 hours starting on day +5
Drug: Mycophenolate mofetil (MMF) — Mycophenolate mofetil 15 mg/kg IV over 2 hours three times a day starting on day +5 will continue until Approximately+35 (+/- two days)
Drug: Cyclophosphamide (Cytoxan) — Cyclophosphamide: 50 mg/kg IV once daily over 2 hours on days +3 and +4, dosed according to ideal body weight

SUMMARY:
Background:

During a transplant, blood stem cells from one person are given to someone else. The cells grow into the different cells that make up the immune system. This can cure people with certain immunodeficiencies. But transplant has many risks and complications.

Objective:

To see if stem cell transplant can be successfully performed in people with primary immunodeficiency disease and cure them.

Eligibility:

People ages 4-69 for whom a primary immunodeficiency (PID) or Primary Immune Regulatory Disorder (PIRD), has caused significant health problems and either standard management has not worked or there are no standard management options, along with their donors

Design:

Donors will be screened under protocol 01-C-0129. They will donate blood or bone marrow.

Participants will be screened with:

Medical history

Physical exam

Blood, urine, and heart tests

CT or PET scans

Before transplant, participants will have dental and eye exams. They will have a bone marrow biopsy. For this, a needle will be inserted through the skin into the pelvis to remove marrow.

Participants will be hospitalized before their transplant. They will have a central catheter put into a vein in their chest or neck. They will get medications through the catheter to prevent complications. Participants will get stem cells through the catheter. They will stay in the hospital for at least 4 weeks. They will give blood, urine, bone marrow, and stool samples. They may need blood transfusions. They may need more scans. They will take more medications.

Participants will have visits on days 30, 60, 100, 180, and 360, and 24 months after the transplant. Then they will have visits once a year for about 5 years

DETAILED DESCRIPTION:
Background:

* With the availability of whole exome sequencing (WES) and whole genome sequencing (WGS) for patients with suspected inborn errors of immunity (IEI), the number of recognized IEI has increased in recent years to over 400 distinct immune defects.
* Allogeneic hematopoietic stem cell transplantation (HSCT) represents a potentially curative therapy for many hematologic diseases.
* Hematopoietic stem cell transplant is now an accepted standard or an appropriate experimental approach for treatment of an increasing number of IEI
* We propose to evaluate the efficacy and safety of allogeneic hematopoietic stem cell transplantation using selected conditioning regimens and selected donor sources in reconstituting normal hematopoiesis and immune function and reversing the disease phenotype in patients with IEI.

Objectives:

-To determine whether allogeneic HSCT in patients with IEI results in sustained donor engraftment defined as neutrophil recovery with ANC >= 500/mm^3 for 3 consecutive days associated with > 50% donor T-cell and myeloid cell donor chimerism by day 100 for diseases characterized by loss of function, and >75% donor T-cell and myeloid cell chimerism for diseases characterized by gain-of-function mutations.

Eligibility:

* Participants ages 4-69 years old with a known IEI, or with clinical evidence of an IEI with a history of recurrent infections requiring prolonged courses of therapy, or evidence of immune dysregulation manifested by autoimmune/autoinflammatory disease, atopy, hemophagocytic lymphohistiocytosis, hypogammaglobulinemia, or impaired response to vaccination. A virally-driven malignancy alone will also constitute a basis for inclusion.
* Have an 8/8, 7/8, or 6/8 HLA-matched related or unrelated donor (HLA -A, -B, -C, DRB1, by high resolution typing) or a haploidentical related donor; unrelated donors are identified through the National Marrow Donor Program.

Design:

For Recipients with Fully Matched Donors

* Patients with IEI receiving a high intensity transplant conditioning regimen will receive a regimen consisting of fludarabine 40 mg/m^2 IV once daily for 4 days on days -6, -5, -4, and -3, busulfan IV once daily for 4 days on days -6, -5, -4, -3 (busulfan dose will be based on pharmacokinetic levels from the test dose or real time pharmacokinetics (PKs) and will be targeted to a daily AUC of 3200-4400 micro Mol min/L (total busulfan exposure of 52-72 mg h/L) (3.2 mg/kg IV per day will be the default dose), and HSCT on day 0.
* Patients with IEI receiving an intermediate intensity transplant conditioning regimen will receive a regimen consisting of fludarabine 40 mg/m2 IV once daily for 4 days on days -6, -5, -4, and -3, busulfan IV once daily for 3 days on days -6, -5, -and -4 (busulfan dose will be based on pharmacokinetic levels from the test dose or real time PKs and will be targeted

to a daily AUC of 3200-4400 micro Mol min/L (total busulfan exposure of 39-54 mg h/L) (3.2 mg/kg IV per day will be the default dose), and HSCT on day 0.

-Patients with IEI receiving a low intensity transplant conditioning regimen will receive a regimen consisting of fludarabine 40 mg/m^2 IV once daily for 4 days on days -6, -5, -4, and -3, busulfan IV once daily for 2 days on days -6, and -5 (busulfan dose will be based on pharmacokinetic levels from the test dose or real time PKs and will be targeted to a daily AUC of 3200-4400 micro Mol min/L (total busulfan exposure of 26-36 mg h/L) (3.2 mg/kg IV per day will be the default dose), and HSCT on day 0.

In all cohorts, alemtuzumab will be given per PI discretion to patients with clinical evidence of immune dysregulation, at the dose of 10 mg/m^2 subcutaneously divided over 3 days, on days -14, -13 and -12.

For Recipients with 7/8 or 6/8 Matched Related or Unrelated Donors and Haploidentical Related Donors

* Patients with IEI receiving a high intensity transplant conditioning regimen will receive a regimen consisting of fludarabine 40 mg/m^2 IV once daily for 4 days on days -6, -5, -4, and -3, busulfan IV once daily for 4 days on days -6, -5, -4, and -3 (busulfan dose will be based on pharmacokinetic levels from the test dose or real time PKs and will be targeted to a daily AUC of 3200-4400 micro Mol min/L (52-72 mg h/L) (3.2 mg/kg IV per day will be the default dose), 200 cGy TBI on day -1, and HSCT on day 0.
* Patients with IEI receiving an intermediate intensity transplant conditioning regimen will receive a regimen consisting of fludarabine 40 mg/m2 IV once daily for 4 days on days - 6, -5, -4, -and 3, busulfan IV once daily for 3 days on days -6, -5, and -4 (busulfan dose will be based on pharmacokinetic levels from the test dose or real time PKs and will be targeted to a daily AUC of 3200-4400 micro Mol min/L (39-54 mg h/L) (3.2 mg/kg IV per day will be the default dose), 200 cGy TBI on day -1, and HSCT on day 0.
* Patients with IEI receiving a low intensity transplant conditioning regimen will receive a regimen consisting of fludarabine 40 mg/m2 IV once daily for 4 days on days -6, -5, -4, and -3, busulfan IV once daily for 2 days on day -6 and -5 (busulfan dose will be based on pharmacokinetic levels from the test dose or real time PKs and will be targeted to a daily AUC of 3200-4400 micro Mol min/L (26-36 mg h/L) (3.2 mg/kg IV per day will be the default dose), 200 cGy TBI on day -1, and HSCT on day 0.

In all cohorts, alemtuzumab will be given per PI discretion to patients with clinical evidence of immune dysregulation, at the dose of 10 mg/m2 subcutaneously divided over 3 days, on days -14, -13 and -12.

For Post-Transplant GVHD Prophylaxis

-Post-transplant GVHD prophylaxis in all groups will consist of cyclophosphamide 50 mg/kg IV once daily for 2 days on days +3 and +4, along with mycophenolate mofetil from day +5 to approximately day +35 and tacrolimus from day +5 to approximately day +180.

If there is no evidence of GVHD, tacrolimus will be stopped or tapered at approximately day +180.

ELIGIBILITY:
* INCLUSION CRITERIAl:
* Age >= 4 years and <=69 yo with Weight >=12 kilograms
* Mutation in a known monogenic (IEI) gene performed by a CLIA certified laboratory, who have failed standard medical management, or when no standard medical management is available.

OR

Patients without a known IEI mutation may be eligible if they have a clinical history that is characteristic of an individual with an immune defect including a history of infections requiring prolonged courses of therapy or evidence of immune dysregulation manifested by autoimmune/autoinflammatory disease, atopy, hemophagocytic lymphohistiocytosis, hypogammaglobulinemia, or impaired response to vaccination. A virally-driven malignancy alone will also constitute basis for inclusion.

* Availability of an 8/8, 7/8, or 6/8 HLA-matched related or unrelated donor (if the mismatch is at DQ this will be considered an 8/8 matched donor), or a haploidentical related donor. Karnofsky or Lansky performance status of >= 40%
* Adequate end-organ function, as measured by:

  --Left ventricular ejection fraction > 40%, preferably by 2-D echocardiogram (ECHO) obtained within 60 days prior to enrollment.
* Creatinine: Adult patients: <= 2.0 mg/dl and creatinine clearance >= 30 ml/min; Pediatric patients (<18 years old): creatinine < 1.5 mg/dL and a creatinine clearance, using the Schwartz Formula > 30 mL/min/1.73m^2.

  * Serum conjugated bilirubin < 2.5 mg/dl; serum ALT and AST <= 5 times upper

limit of normal.

--Pulmonary function tests: FEV1 > 30% and DLCO >30%. Children who are unable to have DLCO assessed due to age, are still eligible if no evidence of dyspnea at rest and no need for supplemental oxygen.

* Ability of subject or parent/guardian to understand and the willingness to sign a written informed consent document. For subjects <18 years old, their legal guardian must give informed consent. Pediatric patients will provide assent.
* As therapeutic agents used in this trial may be harmful to a fetus, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for at least one year post-allo HCT. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in the study, she should inform her treating physician immediately.
* Willingness to remain in the NIH hospital or, if discharged, stay close to the NIH, for a minimum of 100 days after transplant or longer, if there are complications. If outpatient in the first 100 days after transplant, patient must commit to having an adult caregiver with them at all times.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents (with the exception of virus-specific therapy e.g. cytotoxic T-cells for the treatment of viral infection/reactivation prior to allo HCT).
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* HIV-positive patients are ineligible because these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents (steroids, cyclophosphamide, busulfan, tacrolimus, sirolimus, MMF, G-CSF, alemtuzumab) used in the study
* Active psychiatric disorder which is deemed by the PI to have significant risk of compromising compliance with the transplant protocol or which does not allow for appropriate informed consent
* Pregnant women are excluded from this study because the study agents have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study agents, breastfeeding should be discontinued if the mother is treated with the study agents.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 4 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Sustained donor engraftment | baseline to day +100
  neutrophil recovery with ANC >/= 500/mm^3 for 3 consecutive days with >50% or >75% T-cell and myeloid donor chimerism

SECONDARY OUTCOMES:
Reversal of the immunological abnormalities | 1 through 5 years post transplant
  Cumulative correction of disease-specific immunological abnormalities by 1-5 years post transplant
Reversal of the clinical phenotype | 1 and 2 years post transplant
  Cumulative improvement of clinical phenotype consistent with the replacement of hematopoietic cells at 1 -5 years post transplant
regimen-related mortality | +180 and 1 year post transplant
  Cumulative incidence of transplant-related mortality at 180 days and 1 year post transplant
Overall survival | 1 through 5 years post transplant
  Time from transplant to death of any cause
infection and viral reactivation | +180 and 1 year post transplant
  Cumulative incidence of transplant-related mortality at 180 days and 1 year post transplant
Incidence of Chronic Graft-versus-host disease | 1 and 2 years post transplant
  Cumulative incidence of chronic graft versus host disease at 1 and 2 years post transplant
Incidence of Acute Graft-versus-host disease | 100 days post transplant
  Cumulative incidence of acute graft versus host disease at day 100 post transplant
Event free survival | 1 through 5 years post transplant
  Time from transplant to death of any cause, primary or secondary graft failure, or second transplant

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Yun Pai, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Derived] Arnold DE, Kaviany S, Aluri J, Calvo KR, Mehta SS, Tobin JM, Schuettpelz L, Saucier N, Schmitz EG, Murguia-Favela L, Wright NAM, De Ravin SS, Rao VK, Holland SM, Bleesing J, Loughran TP, Feith DJ, Powell J, Ratan A, Warren JT, Pai SY, Bednarski JJ, Connelly JA, Cooper MA. Clinical Characteristics, Management, and Hematopoietic Cell Transplantation of Patients with TLR8 Gain-of-Function. Blood Adv. 2025 Dec 10:bloodadvances.2025016338. doi: 10.1182/bloodadvances.2025016338. Online ahead of print. PMID 41370196
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-C-0070.html